CLINICAL TRIAL: NCT04820478
Title: Efficacy and Tolerability of Beta Hydroxybutyrate Ester in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: KETO-ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Prof., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KETO-ALS V 1.41
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: nutrition; beta hydroxybutyrate ester; high-caloric; ketone ester; ketone monoester
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo-controlled study, using a placebo with similar look and taste in similar bottles; the study is double-blinded, i.e. patients and study personnel are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta Hydroxybutyrate Ester (Experimental): 3 x 10 g beta hydroxybutyrate ester per day, in addition to normal food intake and standard therapy (2 x 50 mg riluzole per day)
  Interventions: Dietary Supplement: Beta Hydroxybutyrate Ester (KetoneAid KE4)
- Placebo (Placebo Comparator): matching placebo, in addition to normal food intake and standard therapy (2 x 50 mg riluzole per day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta Hydroxybutyrate Ester (KetoneAid KE4) — see arm/group description
  Arms: Beta Hydroxybutyrate Ester
Dietary Supplement: Placebo — see arm/group description
  Arms: Placebo

SUMMARY:
Weight loss is a known negative prognostic factor in amyotrophic lateral sclerosis (ALS). One potential mechanism of weight loss in ALS is a disturbance of the mitochondrial complex I which causes an energy deficit in affected cells. Over the last years, various interventional studies targeting the energy deficit in ALS yielded promising results; however,it is still unclear which kind of nutrition or nutritional supplement is most beneficial. Ketone bodies represent a logical therapeutic option in ALS as ketone bodies are an extremely high-energetic substrate which yields the double amount of adenosine triphosphate (ATP) per mole compared to glucose. The human liver is able to synthesize ketone bodies (beta-hydroxybutyrate, acetone, and aceto-acetate) from fat in times of glucose shortage, for example after a prolonged period of fasting. This metabolic shift is the underlying principle of the ketogenic diet, a carbohydrate-free, fat-rich diet which has been successfully tested in other neurodegenerative diseases such as Alzheimer's and Parkinson's disease. In the ALS mouse model, a ketogenic diet was associated with a slower decline of motor function. However, a ketogenic diet is difficult to implement in ALS as it requires a long-term change of eating habits, which is difficult to achieve due to progressive dysphagia, fast worsening of general condition, and limited survival. Therefore, the direct administration of ketone bodies yields a more realistic alternative in ALS as it is easy to apply and allows to maintain the usual eating habits. In this study, we hypothesize that the administration of 3 x 10 g beta hydroxybutyrate ester per day (in addition to normal food intake and the standard medication of 2 x 50 mg riluzole) slows down disease progression as measured by neurofilament light chains (NfL) in serum after 6 months compared to placebo. Power calculation relies on the results of the lipids and calories for ALS (LIPCAL-ALS) study which tested the effect of a high-caloric fatty nutritional supplement in ALS. The study revealed that NfL serum values declined significantly in the intervention group while remaining stable in the placebo group over the course of the study. Assuming a similar effect size for ketone bodies, we calculated that 76 patients had to be included in the current trial.

ELIGIBILITY:
Inclusion Criteria:

* Probable (clinically or laboratory) or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria
* loss of Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) of ≥ 0.33 points per month since onset (first paresis), based on the formula: (48 - score at screening visit) / (months between onset and screening visit)
* age ≥ 18 years
* continuously treated with 100 mg riluzole per day for at least 4 weeks
* capable of thoroughly understanding all information given and giving full informed consent according to good clinical practice (GCP)

Exclusion Criteria:

* hyperinsulinism
* pyruvate decarboxylase deficit
* disturbance of fatty acid oxidation
* disturbance of gluconeogenesis
* acute porphyria
* metabolism disorders which prevent utilization or degradation of ketone bodies
* severe gastro-esophageal reflux
* renal insufficiency (medical history and/or elevated serum creatinine levels and/or glomerular filtration rate (GFR) <90 ml/min
* previous participation in another interventional study within the preceding 4 weeks
* tracheostomy
* pregnancy or breast-feeding females
* evidence of a major psychiatric disorder or clinically evident dementia
* intake of diuretics
* severe dysphagia
* nutrition via percutaneous endoscopic gastrostomy (PEG)
* electrolyte or acid-base imbalance
* heart failure New York Heart Association (NYHA) II or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Neurofilament Light Chain | 6 months
  Neurofilament Light Chain (NfL) serum levels

SECONDARY OUTCOMES:
Survival | 6 months
  Survival (time to death or tracheostomy)
Amyotrophic Lateral Sclerosis Functional Rating Scale Revised | 6 months
  Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) score, measured as individual slope (loss of points per month)
Body Mass Index | 6 months
  Body Mass Index (BMI), weight (in kg) and height (in m) will be combined to report BMI in kg/m^2
Slow Vital Capacity | 6 months
  Slow Vital Capacity (sVC)
Resting Energy Expenditure | 6 months
  Resting Energy Expenditure (REE), measured by indirect calorimetry
Fatt mass | 6 months
  Fat mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Total Body Water | 6 months
  total body water (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Muscle Mass | 6 months
  muscle mass (% of total body mass) measured by bioelectrical impedance analysis (BIA)
Fat Free Mass | 6 months
  fat free mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Body Cell Mass | 6 months
  body cell mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Extracellular Mass | 6 months
  extracellular mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Lean Body Mass | 6 months
  lean body mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Individual Quality of Life | 6 months
  Individual Quality of Life, measured by the Euro Quality of Life (EQ-5D-5L) questionnaire
Neurofilament Phosphorylated Heavy Chain | 6 months
  Neurofilament Phosphorylated Heavy Chain (pNfH) in cerebrospinal fluid (CSF)
Beta Hydroxybutyrate | 6 months
  Beta Hydroxybutyrate serum levels
Acetone | 6 months
  Acetone concentration in urine
Appetite | 6 months
  Appetite, measured by the Council of Appetite Questionnaire (CNAQ)
Eating Habits | 6 months
  Eating Habits, evaluated by the Ulm Nutrition Questionnaire (UNQ; see LIPCAL study)
Adverse Events | 6 months
  Terms and frequencies of Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ulm, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification as well as the study protocol will be available. Data will be available beginning 3 months and ending 5 years following article publication. Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims provided in the approved proposal. Proposals should be directed to johannes.dorst@uni-ulm.de; to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: 3 months to 5 years following article publication
Access Criteria: Data will be shard for analyses to achieve the aims provided in the approved proposal. Proposals should be directed to johannes.dorst@uni-ulm.de; to gain access, data requestors will need to sign a data access agreement.
URL: https://www.uniklinik-ulm.de/neurologie.html

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Dupuis L, Oudart H, Rene F, Gonzalez de Aguilar JL, Loeffler JP. Evidence for defective energy homeostasis in amyotrophic lateral sclerosis: benefit of a high-energy diet in a transgenic mouse model. Proc Natl Acad Sci U S A. 2004 Jul 27;101(30):11159-64. doi: 10.1073/pnas.0402026101. Epub 2004 Jul 19. PMID 15263088
- [Background] Desport JC, Preux PM, Truong TC, Vallat JM, Sautereau D, Couratier P. Nutritional status is a prognostic factor for survival in ALS patients. Neurology. 1999 Sep 22;53(5):1059-63. doi: 10.1212/wnl.53.5.1059. PMID 10496266
- [Background] Desport JC, Preux PM, Magy L, Boirie Y, Vallat JM, Beaufrere B, Couratier P. Factors correlated with hypermetabolism in patients with amyotrophic lateral sclerosis. Am J Clin Nutr. 2001 Sep;74(3):328-34. doi: 10.1093/ajcn/74.3.328. PMID 11522556
- [Background] Dorst J, Cypionka J, Ludolph AC. High-caloric food supplements in the treatment of amyotrophic lateral sclerosis: a prospective interventional study. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Dec;14(7-8):533-6. doi: 10.3109/21678421.2013.823999. Epub 2013 Aug 14. PMID 23944684
- [Background] Wills AM, Hubbard J, Macklin EA, Glass J, Tandan R, Simpson EP, Brooks B, Gelinas D, Mitsumoto H, Mozaffar T, Hanes GP, Ladha SS, Heiman-Patterson T, Katz J, Lou JS, Mahoney K, Grasso D, Lawson R, Yu H, Cudkowicz M; MDA Clinical Research Network. Hypercaloric enteral nutrition in patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet. 2014 Jun 14;383(9934):2065-2072. doi: 10.1016/S0140-6736(14)60222-1. Epub 2014 Feb 28. PMID 24582471
- [Background] Dorst J, Schuster J, Dreyhaupt J, Witzel S, Weishaupt JH, Kassubek J, Weiland U, Petri S, Meyer T, Grehl T, Hermann A, Jordan B, Grosskreutz J, Zeller D, Boentert M, Schrank B, Prudlo J, Winkler AS, Gorbulev S, Roselli F, Dupuis L, Otto M, Ludolph AC. Effect of high-caloric nutrition on serum neurofilament light chain levels in amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2020 Sep;91(9):1007-1009. doi: 10.1136/jnnp-2020-323372. Epub 2020 Aug 11. No abstract available. PMID 32788256
- [Background] Steinacker P, Feneberg E, Weishaupt J, Brettschneider J, Tumani H, Andersen PM, von Arnim CA, Bohm S, Kassubek J, Kubisch C, Lule D, Muller HP, Muche R, Pinkhardt E, Oeckl P, Rosenbohm A, Anderl-Straub S, Volk AE, Weydt P, Ludolph AC, Otto M. Neurofilaments in the diagnosis of motoneuron diseases: a prospective study on 455 patients. J Neurol Neurosurg Psychiatry. 2016 Jan;87(1):12-20. doi: 10.1136/jnnp-2015-311387. Epub 2015 Aug 21. PMID 26296871
- [Background] Grammatikopoulou MG, Goulis DG, Gkiouras K, Theodoridis X, Gkouskou KK, Evangeliou A, Dardiotis E, Bogdanos DP. To Keto or Not to Keto? A Systematic Review of Randomized Controlled Trials Assessing the Effects of Ketogenic Therapy on Alzheimer Disease. Adv Nutr. 2020 Nov 16;11(6):1583-1602. doi: 10.1093/advances/nmaa073. PMID 32597927
- [Background] Phillips MCL, Murtagh DKJ, Gilbertson LJ, Asztely FJS, Lynch CDP. Low-fat versus ketogenic diet in Parkinson's disease: A pilot randomized controlled trial. Mov Disord. 2018 Aug;33(8):1306-1314. doi: 10.1002/mds.27390. Epub 2018 Aug 11. PMID 30098269
- [Background] Zhao Z, Lange DJ, Voustianiouk A, MacGrogan D, Ho L, Suh J, Humala N, Thiyagarajan M, Wang J, Pasinetti GM. A ketogenic diet as a potential novel therapeutic intervention in amyotrophic lateral sclerosis. BMC Neurosci. 2006 Apr 3;7:29. doi: 10.1186/1471-2202-7-29. PMID 16584562
- [Background] Clarke K, Tchabanenko K, Pawlosky R, Carter E, Todd King M, Musa-Veloso K, Ho M, Roberts A, Robertson J, Vanitallie TB, Veech RL. Kinetics, safety and tolerability of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate in healthy adult subjects. Regul Toxicol Pharmacol. 2012 Aug;63(3):401-8. doi: 10.1016/j.yrtph.2012.04.008. Epub 2012 May 3. PMID 22561291
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194
- [Background] Poffe C, Ramaekers M, Van Thienen R, Hespel P. Ketone ester supplementation blunts overreaching symptoms during endurance training overload. J Physiol. 2019 Jun;597(12):3009-3027. doi: 10.1113/JP277831. Epub 2019 May 22. PMID 31039280
- [Background] Hashim SA, VanItallie TB. Ketone body therapy: from the ketogenic diet to the oral administration of ketone ester. J Lipid Res. 2014 Sep;55(9):1818-26. doi: 10.1194/jlr.R046599. Epub 2014 Mar 5. PMID 24598140